CLINICAL TRIAL: NCT02936232
Title: Severe Sepsis and Septic Shock Registry
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other); Hallym University Kangnam Sacred Heart Hospital (Other); Gangnam Severance Hospital (Other); Kyungpook National University Hospital (Other); Kyunghee University Medical Center (Other); Korea University Guro Hospital (Other); Korea University Anam Hospital (Other); The Catholic University of Korea (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Severance Hospital (Other); Ulsan University Hospital (Other); Inje University Ilsan Paik Hospital (Other); Chonnam National University Hospital (Other); Chonbuk National University Hospital (Other); Jeju National University Hospital (Other); Chosun University Hospital (Other); Hallym University Medical Center (Other); Hanyang University Seoul Hospital (Other); Bucheon St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Gil Joon Suh, Professor, Seoul National University Hospital
Other Study IDs: 1408-003-599
Record Dates: First submitted 2016-10-09; First posted 2016-10-18 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to construct multi-center sepsis registry that can be used for data warehousing and clinical research.

DETAILED DESCRIPTION:
This registry prospectively enrolls adult patients with severe sepsis or septic shock in 21 tertiary hospital emergency departments.

Registered data can be used for quality control and clinical research to reduce sepsis-related mortality.

ELIGIBILITY:
Inclusion Criteria:

* two of more systemic inflammatory reaction syndrome criteria fever > 38.3 'C or hypothermia < 36'C, tachycardia over 90 bpm tachypnea over 20 per minute, leukocytosis (WBC over 12k/microL) or leukopenia (WBC below 4k/microL)
* suspected or proven infection
* any organ dysfunction as follows:

  1. cardiovascular (hypotension, systolic blood pressure <90 mmHg, mean arterial pressure <70mmHg)
  2. tissue hypoperfusion (lactate above upper limits laboratory normal)
  3. acute lung injury (PaO2/inspired oxygen fraction < 250 in the absence of pneumonia, PaO2/inspired oxygen fraction < 200 in the presence of pneumonia)
  4. acute kidney injury (Urine output < 0.5mL/kg/hr for at least 2 hrs Serum creatinine > 2.0 mg/dL)
  5. acute liver injury (Total bilirubin > 2mg/dL)
  6. acute coagulopathy (Platelet count < 100,000/μL or prothrombin time, international normalized ratio > 1.5)

Exclusion Criteria:

* age less than 18 years old
* patients with cardiac arrest at presentation
* patients with advanced directives not to deliver aggressive organ supportive management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-08; Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28-day
  According to hospital discharge record review and telephone follow-up.

SECONDARY OUTCOMES:
90-day mortality | 90-day
  According to hospital discharge record review and telephone follow-up.
Organ support treatment (mechanical ventilation) | hospital discharge (non-survivors) or 90 days (survivors)
  According to hospital record review
Organ support treatment (renal replacement therapy) | hospital discharge (non-survivors) or 90 days (survivors)
  According to hospital record review
ICU length of stay | hospital discharge (non-survivors) or 90 days (survivors)
  According to hospital record review
Hospital length of stay | hospital discharge (non-survivors) or 90 days (survivors)
  According to hospital record review

CONTACTS AND LOCATIONS:
Overall Officials: Gil Joon Suh, MD, PhD, Study Director — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Government-Seoul National University Boramae Medical Center, Seoul